CLINICAL TRIAL: NCT00924118
Title: A Safety and Efficacy Evaluation of Sodium Nitrite Injection for the Prevention of Ischemia-Reperfusion Injury Associated With Acute Myocardial Infarction.
Brief Title: Sodium Nitrite in Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Hope Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00023049
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Reperfusion injury; Nitric oxide
MeSH Terms: conditions — Reperfusion Injury | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Nitrite (Experimental): Dose escalation of sodium nitrite.
  Interventions: Drug: Sodium Nitrite
- Open Control (No Intervention): Standard therapy

INTERVENTIONS:
Drug: Sodium Nitrite — Subjects assigned to sodium nitrite will receive an initial infusion of 6 nmol/min/kg for 48 hours. After the first six subjects have been enrolled (3 active drug, 3 control) and if there are no dose limiting toxicities, additional cohorts of six subjects each will be randomized to escalating doses of sodium nitrite versus control for a total of 30 subjects.
  Arms: Sodium Nitrite

SUMMARY:
The purpose of this study is to determine whether the intravenous infusion of sodium nitrite safely prevents ischemia-reperfusion injury in subjects with acute myocardial infarction resulting in improved left ventricular function.

DETAILED DESCRIPTION:
Despite reperfusion therapies, significant myocardial injury continues to occur from ischemic-reperfusion injury. Studies in animal models of acute myocardial infarction suggest that an infusion of sodium nitrite, which is nonenzymatically converted to nitric oxide in the setting of ischemia, significantly reduces ischemia-reperfusion injury resulting in smaller infarcts and improved left ventricular function. The objectives of this phase 2 trial are to determine the tolerability and safety of a 48-hour infusion of sodium nitrite in patients with an acute ST-segment elevation myocardial infarction receiving percutaneous coronary intervention. The efficacy of a 48-hour infusion of sodium nitrite will be determined by noninvasive imaging to determine infarct size and left ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Acute ST segment elevation myocardial infarction
* Eligible for percutaneous coronary intervention

Exclusion Criteria:

* Cardiogenic shock
* Cardiac arrest
* Prior infarct in the infarct related artery
* Hemoglobinopathy, Glucose-6 Phosphate Dehydrogenase (G6PD) deficiency

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Schulman, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez FM, Shiva S, Vincent PS, Ringwood LA, Hsu LY, Hon YY, Aletras AH, Cannon RO 3rd, Gladwin MT, Arai AE. Nitrite anion provides potent cytoprotective and antiapoptotic effects as adjunctive therapy to reperfusion for acute myocardial infarction. Circulation. 2008 Jun 10;117(23):2986-94. doi: 10.1161/CIRCULATIONAHA.107.748814. Epub 2008 Jun 2. PMID 18519850
- [Background] Duranski MR, Greer JJ, Dejam A, Jaganmohan S, Hogg N, Langston W, Patel RP, Yet SF, Wang X, Kevil CG, Gladwin MT, Lefer DJ. Cytoprotective effects of nitrite during in vivo ischemia-reperfusion of the heart and liver. J Clin Invest. 2005 May;115(5):1232-40. doi: 10.1172/JCI22493. Epub 2005 Apr 14. PMID 15841216
- [Background] Rassaf T, Flogel U, Drexhage C, Hendgen-Cotta U, Kelm M, Schrader J. Nitrite reductase function of deoxymyoglobin: oxygen sensor and regulator of cardiac energetics and function. Circ Res. 2007 Jun 22;100(12):1749-54. doi: 10.1161/CIRCRESAHA.107.152488. Epub 2007 May 10. PMID 17495223

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Control: Subjects randomized to open control will receive no experimental therapy.
Period: Overall Study
Arm/Group | Sodium Nitrite | Open Control
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Nitrite | Open Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 59.6 [44 to 76] | 59.2 [46 to 72] | 59.4 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 11 | 14 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Ischemia Area at Risk as Determined by Paired Single-photon Computed Tomography Studies With Technetium Tc99m Sestamibi.
Description: Measured as percentage of left ventricle
Time Frame: 4-5 days from enrollment
Population: Sestamibi imaging proved impossible to obtain emergently and therefore no data was collected.
Arm/Group | Sodium Nitrite | Open Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Left Ventricular Infarct Size
Description: Left ventricular infarct size by Magnetic Resonance Imaging (MRI). Calculated percentage of the left ventricular mass by MRI that has undergone infarction.
Time Frame: 4-5 days following enrollment
Population: Only 2 participants from each arm underwent MRI imaging. Too few subjects underwent MRI imaging to make a statistical comparison. Only those where data was obtained has been reported.
Measure: Mean (Full Range); unit: infarct percentage of left ventricle
Arm/Group | Sodium Nitrite | Open Control
Number analyzed (Participants) | 2 | 2
infarct percentage of left ventricle | 15.5 [7 to 17] | 24 [17 to 31]

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | Sodium Nitrite | Open Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Nitrite (N=15) | Open Control (N=15)
Hypotension (Cardiac disorders) | 4 (4) | 0 (0) — Transient hypotension developed in 4 subjects.
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Two subjects developed nausea during study drug infusion.

LIMITATIONS AND CAVEATS:
The primary and secondary outcomes of this study were limited by too few subjects undergoing these studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes